CLINICAL TRIAL: NCT00332410
Title: Intravenous Voriconazole in Patients With Renal Compromise
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB#0605055
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2015-12

CONDITIONS: Renal Transplant
Keywords: Voriconazole; renal transplant; kidney function; kidneys

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether patients with compromised renal function (CrCl < 50mL/min) receiving intravenous voriconazole experienced any adverse effects related to serum chemistries or other imaging studies of the kidney due to the potential accumulation of the vehicle cyclodextran.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether patients with compromised renal function (CrCl < 50mL/min) receiving intravenous voriconazole experienced any adverse effects related to serum chemistries or other imaging studies of the kidney due to the potential accumulation of the vehicle cyclodextran. t has been previously shown by a large multi-centered, prospective, randomized study that voriconazole is superior to the then gold standard amphotericin B in the treatment of patients with invasive aspergillosis - a disease with significant morbidity and mortality. In patients with these infections who have severe renal insufficiency may be denied the best therapy due to the accumulation of a diluent with unknown clinical consequences. Qualifying and or quantifying these consequences are important to these patients so that potentially life-threatening therapy should not be unduly denied.

ELIGIBILITY:
Inclusion Criteria:

- Patients > 18 years old receiving voriconazole with a serum creatinine of > 2mg/dl (a proxy marker for Creatinine clearance < 50ml/min). Control group in this study will have serum creatinine < 1.5mg/dl. Solid organ transplant patient. Patient that received at least 2 doses of voriconazole.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: solid organ transplant receiving voriconazole with serum creatinine level >2
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2006-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Potoski, Pharm D, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States